CLINICAL TRIAL: NCT06201351
Title: Study of Adaptive Radiotherapy for High-grade Glioma Based on Interfraction Magnetic Resonance Imaging (MRI)
Brief Title: Study of Adaptive Radiotherapy for High-grade Glioma Based on Interfraction MRI
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ping Ai, Clinical Professor, West China Hospital
Other Study IDs: Trial No. 1460, 2023
Record Dates: First submitted 2023-11-28; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: High-grade Glioma
Keywords: adaptive radiotherapy; high-grade glioma; MRI image
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Adaptive radiotherapy group: MRI was performed and adaptive radiotherapy was administered at farction10 and fraction 20 during radiotherapy.
  Interventions: Device: adaptive radiotherapy

INTERVENTIONS:
Device: adaptive radiotherapy — MRI was performed and adaptive radiotherapy was administered at farction10 and fraction 20 during radiotherapy.
  Other Names: ART

SUMMARY:
The changes of target and organs at risk in patients with high-grade glioma during concurrent chemoradiotherapy were evaluated by MRI image between radiotherapy fractions.

DETAILED DESCRIPTION:
To prospectively evaluate the changes of target organs and risk organs in patients with high-grade glioma during concurrent chemoradiotherapy.The related factors causing this change are discussed.The relationship between changes and patient survival was analyzed.A predictive model was established to provide individualized adaptive radiotherapy for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. High-grade glioma was confirmed by pathology after surgery;
3. ECOG score 0-2 points;
4. Receiving the standard STUPP regimen (i.e. 6 weeks of temozolomide concurrent chemoradiotherapy +6 cycles of temozolomide adjuvant chemotherapy);
5. Baseline data available.

Exclusion Criteria:

1. The pathological diagnosis is not clear;
2. No synchronous chemotherapy/adjuvant chemotherapy < 6 cycles;
3. There are other malignant tumors;
4. Previously radiotherapy to the head;
5. Interruption of radiotherapy for more than 5 days;
6. Failure to collect baseline data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-grade glioma confirmed by pathology in our hospital and treated with standard STUPP regimen.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Homogeneity index | up to 2 weeks
  HI: Homogeneity index. Dosimetric change
conformity index | up to 2 weeks
  CI: conformity index. Dosimetric change
Anatomic change | up to 2 weeks
  Dmax Volume

SECONDARY OUTCOMES:
progression-free survival (PFS) | assessed up to 12 months
  progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided